CLINICAL TRIAL: NCT01970579
Title: Clinical Trial on Peripheral Arteries Treated With SeQuent® Please P Paclitaxel Coated Balloon Catheter
Acronym: ConSeQuent
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAG-G-H-1214
Record Dates: First submitted 2013-10-23; First posted 2013-10-28 (Estimated); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Stenosis; Restenosis
MeSH Terms: conditions — Constriction, Pathologic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paclitaxel coated balloon (Experimental)
  Interventions: Device: Paclitaxel coated balloon
- uncoated PTA catheter (Active Comparator)
  Interventions: Device: uncoated PTA catheter

INTERVENTIONS:
Device: Paclitaxel coated balloon — * Treatment of target lesion with study balloon (coated). Diameter of treatment balloon = RVD
  * Each study balloon must only be used once (except postdilatation is necessary which may be done with the same balloon used for the initial dilatation)
  * Treatment balloon must be 20 mm longer than lesion length (to assure balloon overlap of 10 mm proximal and distal to lesion)
  * If two treatment balloons are necessary overlap between the balloon must be 10 mm
  * Inflation pressure 7-10 atm
  * Intraluminal defects or haziness should be treated with additional inflations and/or aggressive anti-platelet agents or bailout stenting
  Other Names: SeQuent® Please P; Drug coated balloon
  Arms: Paclitaxel coated balloon
Device: uncoated PTA catheter — * Treatment of target lesion with study balloon (uncoated). Diameter of treatment balloon = RVD
  * Each study balloon must only be used once (except postdilatation is necessary which may be done with the same balloon used for the initial dilatation)
  * Treatment balloon must be 20 mm longer than lesion length (to assure balloon overlap of 10 mm proximal and distal to lesion)
  * If two treatment balloons are necessary overlap between the balloon must be 10 mm
  * Inflation pressure 7-10 atm
  * Intraluminal defects or haziness should be treated with additional inflations and/or aggressive anti-platelet agents or bailout stenting.
  Other Names: POBA
  Arms: uncoated PTA catheter

SUMMARY:
The aim of the study is to assess the safety and efficacy of the paclitaxelreleasing balloon catheter SeQuent® Please P to treat de novo and restenotic lesions in the superficial femoral artery and the proximal two segments of the popliteal artery with reference diameters ≥ 4mm & ≤ 7mm and lesion lengths ≥ 4 cm & ≤ 27 cm. It is the intention of this trial to treat suitable target lesions with DCB only.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to treat the target lesion according to the DCB only concept
* Patients in Rutherford classes 2 through 4 (corresponding to Fontaine stage IIb to III)
* Patients eligible for peripheral revascularization by means of PTA
* Patients must be ≥ 18 years of age
* Patients who are mentally and linguistically able to understand the aim of the study and to show sufficient compliance in following the study protocol
* Patients must agree to undergo the 6-month angiographic and clinical follow-up
* Patients must agree to undergo the 1 and 2 year clinical follow-up
* Patient is able to verbally acknowledge an understanding of the associated risks, benefits, and treatment alternatives to therapeutic options of this trial. The patients, by providing their informed consent, agree to these risks and benefits as stated in the patient informed consent document.
* Peripheral lesions in the native SFA or popliteal artery with reference vessel diameters between ≥ 4.0 and ≤ 7.0 mm, lesions lengths ≥ 4 cm and ≤ 27 cm as angiographically documented
* Diameter stenosis pre-procedure must be ≥ 70%
* Target lesion in the SFA or popliteal artery (first two proximal segments)*.

  * as far as applicable distance of the target lesion to a previously implanted stent should be about 1cm
* Vessels must have adequate runoff with at least one vessel to the foot.
* Treatment of max. two lesions is permitted.

Exclusion Criteria:

* Patients with Rutherford class 5 or 6
* Women who are known or suspected to be pregnant. Hence, patients will be advised to use an adequate birth control method up to and including the 6-month follow-up.
* Patients with an expected life span of less than 24 months
* Patients with bleeding diathesis in whom anticoagulation or anti-platelet medication is contraindicated
* Patients who had a cerebral stroke < 6 months prior to the procedure
* Patients with unstable angina pectoris
* Patients with acute myocardial infarction within the past 2 weeks
* Patient participates in other clinical trials involving any investigational device or drug that interfere with the effects to be studied in this trial.
* Interventional treatment at the contralateral leg within 2 weeks prior to or after the study intervention
* Untreated hyperthyroidism
* Patient has presence or history of severe renal failure (GFR < 30ml/min) and is therefore not eligible for angiography.
* Post transplantation of any organ or immune suppressive medication
* Other disease to jeopardize follow-up (e.g. malignoma)
* Addiction to any drug or to alcohol (WHO definition)
* Patients with clinically significant aneurysmal disease of the popliteal, femoral or iliac artery and patients with history of clinically significant abdominal aortic aneurysm
* Patients with any type of surgical/interventional procedures within 4 weeks prior to or planned after study intervention (if those may interfere with the peripheral study intervention and/or patient's ability to perform the follow up examinations)
* Conditions which prevent the intake of the double anti-platelet therapy for two months
* Patients with contraindication for drug-eluting balloon angioplasty given in the instruction for use
* Patients under administrative or judicial custody (§20 Act on Medical Devices, Germany)
* Strongly calcified lesions with circumferential presence of calcifications and a lesion length of > 4 cm
* Chronic total occlusions longer than 10 cm
* Lesion below the knee requiring treatment
* Target lesion within a bypass graft
* In-stent restenosis
* Lesions treated with DCB
* Concomitant use of atherectomy, cryoplasty or laser therapy
* Inflow lesion (proximal to the study lesion) with flow limitation not being successfully treated prior to the study lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Late Lumen Loss | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Albrecht, MD, Principal Investigator — Vivantes Klinikum Neukölln, Berlin, Germany
Locations (7):
- Germany (7):
  - Universitäts-Herzzentrum Freiburg Bad Krozingen, Bad Krozingen
  - Vivantes Klinikum Neukölln, Berlin
  - Ev. Krankenhaus Hubertus, Berlin
  - Klinikum der Otto-von-Guericke-Universität Magdeburg, Magdeburg
  - Klinikum Magdeburg, Magdeburg
  - Deutsches Herzzentrum München, München
  - RoMed Klinikum Rosenheim, Rosenheim

REFERENCES:
- [Derived] Albrecht T, Waliszewski M, Roca C, Redlich U, Tautenhahn J, Pech M, Halloul Z, Gogebakan O, Meyer DR, Gemeinhardt I, Zeller T, Muller-Hulsbeck S, Ott I, Tepe G. Two-Year Clinical Outcomes of the CONSEQUENT Trial: Can Femoropopliteal Lesions be Treated with Sustainable Clinical Results that are Economically Sound? Cardiovasc Intervent Radiol. 2018 Jul;41(7):1008-1014. doi: 10.1007/s00270-018-1940-1. Epub 2018 Mar 27. PMID 29589098
- [Derived] Tepe G, Gogebakan O, Redlich U, Tautenhahn J, Ricke J, Halloul Z, Meyer DR, Waliszewski M, Schnorr B, Zeller T, Muller-Hulsbeck S, Ott I, Albrecht T. Angiographic and Clinical Outcomes After Treatment of Femoro-Popliteal Lesions with a Novel Paclitaxel-Matrix-Coated Balloon Catheter. Cardiovasc Intervent Radiol. 2017 Oct;40(10):1535-1544. doi: 10.1007/s00270-017-1713-2. Epub 2017 Jun 28. PMID 28660441